CLINICAL TRIAL: NCT06430957
Title: Evaluation of OSA Risk Levels in the Preoperative Period of Adult Patients With Planned Dental Procedures Under Anesthesia and Correlation With Postoperative Complications; A Multicenter Study
Brief Title: OSA Risk Level in Dental Patients and Correlation With Complications After General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gözde Nur Erkan, Assistant Professor Doctor, Medical Doctor, Kırıkkale University
Other Study IDs: KU-ERKAN-002
Record Dates: First submitted 2024-05-14; First posted 2024-05-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea Risk Management; Postoperative Complications; Dental Caries Under General Anesthesia; Obstructive Sleep Apnea of Adult
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Group lowSTOP-B: Study group including patients in the low-risk group in the assessment to be made with STOP-BANG questionnaire.
  Interventions: Other: The STOP-BANG questionnaire for determining OSA risk level.; Other: Record of postoperative complications
- Group intermediateSTOP-B: Study group including patients in the medium-risk group in the assessment to be made with STOP-BANG questionnaire.
  Interventions: Other: The STOP-BANG questionnaire for determining OSA risk level.; Other: Record of postoperative complications
- Group highSTOP-B: Study group including patients in the high-risk group in the assessment to be made with STOP-BANG questionnaire.
  Interventions: Other: The STOP-BANG questionnaire for determining OSA risk level.; Other: Record of postoperative complications
- Group noneASA: The study group that includes patients who are not at risk for OSA in the evaluation with the criteria recommended by the ASA.
  Interventions: Other: ASA recommended criteria for determining OSA risk level.; Other: Record of postoperative complications
- Group mildASA: Study group including patients in the mild-risk group for OSA in the evaluation with the criteria recommended by the ASA.
  Interventions: Other: ASA recommended criteria for determining OSA risk level.; Other: Record of postoperative complications
- Group moderateASA: Study group including patients in the moderate-risk group for OSA in the evaluation with the criteria recommended by the ASA.
  Interventions: Other: ASA recommended criteria for determining OSA risk level.; Other: Record of postoperative complications
- Group severeASA: Study group including patients in the severe-risk group for OSA in the evaluation with the criteria recommended by the ASA.
  Interventions: Other: ASA recommended criteria for determining OSA risk level.; Other: Record of postoperative complications

INTERVENTIONS:
Other: The STOP-BANG questionnaire for determining OSA risk level. — An assessment questionnaire including OSA-related physical characteristics and symptoms and signs to be questioned individually in each patient will be examined by the physician.
  Groups: Group highSTOP-B; Group intermediateSTOP-B; Group lowSTOP-B
Other: ASA recommended criteria for determining OSA risk level. — An assessment questionnaire including OSA-related physical characteristics and symptoms and signs to be questioned individually in each patient will be examined by the physician.
  Groups: Group mildASA; Group moderateASA; Group noneASA; Group severeASA
Other: Record of postoperative complications — Respiratory complications as laryngospasm/bronchospasm, apnea, hypoxia, duration and amount of need for additional oxygen support and recovery time (duration of modified aldrete score of 9 and above) will be recorded.

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep-related respiratory dysfunction. The prevalence of OSA is increasing with the increasing rates of obesity and elderly population worldwide. Perioperative anesthesia management should be adjusted to improve patient safety in patients with OSA. In OSA patients, positive pressure ventilation support may be required in the preoperative period, various ventilation strategies may be required in the intraoperative period, different pharmacologic agents may need to be avoided, and intensive care unit follow-up or noninvasive ventilation support may be required in the postoperative period. However, it is reported that a significant percentage of OSA patients remain undiagnosed. ASA (American Society of Anesthesiologists) has reported the criteria that should be questioned in order to determine the risk of patients in terms of OSA and to initiate the diagnostic process in risky patients and to make appropriate anesthesiologic arrangements in the perioperative period. In addition, the STOP-BANG assessment scale, which is widely used all over the world in OSA risk assessment, is also used in OSA risk assessment. It is thought that dental caries and extraction needs may be higher in OSA patients, especially since open-mouth sleeping accompanies the situation. In this respect, it is also important for patients to be diagnosed with OSA as it may prevent dental damage due to open-mouth sleeping in the future. Identifying patients at risk for OSA and directing them to the diagnostic process is very important for patient safety. Within the scope of the study, the criteria recommended by ASA and STOP-BANG score will be evaluated and recorded. Risk stratification in terms of STOP-BANG questionnaire and ASA criteria will be done separately for each patient and for each classification method. Patients at high risk will be consulted to the relevant medical department in the preoperative period for further investigation and treatment. In addition, it is aimed to correlate the risk levels determined in the study with postoperative respiratory complications and recovery time.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-80 years of age who apply to the anesthesia clinic for dental procedures planned to be performed under general anesthesia
* Patients without a previous diagnosis of OSA

Exclusion Criteria:

* Individuals who do not want to participate in the study
* Patients previously diagnosed with OSA
* Necessity of emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-80 years who applied to the anesthesia clinic for dental procedures planned to be performed under general anesthesia and who had no previous diagnosis of OSA.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Determination of OSA risk levels of patients | Preoperative period
  The STOP-BANG questionnaire and the criteria recommended by the ASA, which are recommended to be used routinely worldwide to determine OSA risk level, will be questioned in each patient. Patients with moderate and high risk scores from the STOP-BANG questionnaire and patients with significant OSA risk level according to ASA criteria will be referred to the pulmonology department and further evaluation will be requested. If deemed necessary by the Pulmonology department, a sleep test will be performed. With the sleep test result, the OSA risk level of the patients will be classified as none, mild, moderate and severe in terms of ASA criteria.
Postoperative respiratory complications | For 4 hours after the end of surgery
  Respiratory complications including laryngospasm/bronchospasm, apnea, hypoxia that may develop in the postoperative period in patients, the duration of the need for additional oxygen support above the expected duration will be observed and recorded.
Follow-up of indicators of airway obstruction | For 4 hours after the end of surgery
  As indicators of airway obstruction; snoring/whistling respiration, hypertension and intercostal/sternal retractions will be observed and recorded in the study follow-up form.
Duration of recovery | For 30 minutes after the end of surgery
  Duration of recovery (modified aldrete score of 9 and above) will be recorded

SECONDARY OUTCOMES:
Comparison of the effectiveness of STOP-BANG questionnaire and ASA criteria in determining OSA risk level | Perioperative period
  Patients who will receive an intermediate or high risk score from either of the two assessment questionnaires will be referred for further evaluation and diagnosis of suspected OSA. At the end of the diagnostic process, it is planned to investigate which of the two scoring systems more successfully identifies patients with OSA and assigns a higher risk.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University Faculty of Dentistry, Kayseri
  - Kırıkkale University Faculty of Dentistry, Kırıkkale

IPD SHARING:
Plan to Share IPD: Undecided